CLINICAL TRIAL: NCT03476122
Title: Application of an Automated Liquid Biopsy System in the Detection of Colorectal Cancer
Brief Title: Clinical Application of an Automated Liquid Biopsy Platform for Early Detection of Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CellMaxLife (Industry)
Responsible Party: Sponsor
Other Study IDs: CMx-CTC-CRC-001
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Colo-rectal Cancer
Keywords: Colorectal cancer; CRC; Circulating tumor cells; CTCs; Early detection; Automated
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Group: The disease group is diagnosed with colorectal cancer 0-4 and has not been treated.
- Control Group: The control group will receive Colonoscopy

SUMMARY:
Colorectal cancer (CRC) is among the most preventable cancers when precancerous lesions are detected at an early stage. Current screening methods for CRC require bowel prep or stool-based testing that are inconvenient, resulting in low compliance. Stool based tests have limited sensitivity for the detection of precancerous lesions.

The CMx platform has been showed to be able to the detection of Circulating Tumor Cells (CTCs) in high sensitivity and specificity. In published studies, circulating Tumor Cells (CTCs) are captured and quantified in advanced-stages of colorectal cancer. In order to detect early and pre-cancer circulating tumor cells, we have developed an Automated Liquid Biopsy Platform that improves the detection of CTCs in early cancer stages. Therefore, this study goals are: 1) to establish a standard detection process utilizing the Automated Liquid Biopsy Platform. 2) Parallel comparison of laboratory manual operation and Automated Liquid Biopsy Platform. 3) Verify the feasibility of use of an Automated Liquid Biopsy Platform in the clinical setting.

DETAILED DESCRIPTION:
1. Selection of patients:

   A. The disease group includes 300 patients diagnosed with stages 0-4 colorectal cancer not previously treated.

   B. The control group includes 450 control subjects who will undergo a colonoscopy procedure.
2. Study stages

   Stage I: The laboratory manually analyzes circulating tumor cells to establish a standard detection process for Automated Liquid Biopsy System

   Stage II: Comparison analysis between manual and Automated Liquid Biopsy Platform, establishing the procedural and analytical models for the Automated Liquid Biopsy Platform

   Stage III: Verification of the feasibility of use of an Automated Liquid Biopsy Platform in the clinical setting.
3. Methods

I. CTC isolation Peripheral blood drawn from subjects will be processed using the CMx platform or the automated liquid biopsy system for detection and capture.

II. Characterization of isolated CTC using Immunofluorescence Staining

III. CRC-related gene expression The serum and circulating tumor cells isolated from the blood will be used to extract RNA, and then be analyzed with the expression of different genes by real-time quantitative polymerase chain reaction (real-time PCR).

ELIGIBILITY:
Inclusion Criteria:

* 1. The disease group is diagnosed with colorectal cancer 0-4 and has not been treated.
* 2. The control group will receive Colonoscopy
* 3. Above 20 years old

Exclusion Criteria:

* 1. Refuse to sign the informed consent form
* 2. Received surgery within one month
* 3. Previous cancer history
* 4. Autoimmune diseases
* 5. Chronic inflammatory diseases
* 6. Acute inflammatory or infectious diseases in three months
* 7. Myelodysplastic syndromes and myeloproliferative disorder
* 8. Other diseases decided by PI

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2021-03-13 (Estimated)

PRIMARY OUTCOMES:
Detection of circulating tumor cells | Prior to treatment or colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Sy Tsai, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan